CLINICAL TRIAL: NCT05307835
Title: Clinical Study of a Personalized Neoantigen Vaccine in Esophagus Cancer Patients Who Have Completed Adjuvant Therapy Following Neoadjuvant Therapy and Surgical Resection
Brief Title: Neoantigen Vaccine in Esophagus Cancer Patients Following Neoadjuvant Therapy and Surgical Resection
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Hangzhou Neoantigen Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INEO-P-006
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Resectable Esophageal Cancer
Keywords: has received neoadjuvant therapy; At high risk of recurrence
MeSH Terms: interventions — Granulocyte-Macrophage Colony-Stimulating Factor; Adjuvants, Immunologic; Colony-Stimulating Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalized neoantigen vaccines (Experimental): iNeo-Vac-P01 (peptides)： 300 mcg per peptide
  Interventions: Biological: iNeo-Vac-P01; Biological: GM-CSF

INTERVENTIONS:
Biological: iNeo-Vac-P01 — iNeo-Vac-P01 (peptides)： 4 x 300 mcg per peptide given on days 1, 4, 8, 15, 22, 52, and 82 for a total of 7 doses;
  Other Names: Neoantigen peptides
Biological: GM-CSF — 4 x 40 mcg (total dose 160 mcg) given on days 1, 4, 8, 15, 22, 52, and 82 for a total of 7 doses
  Other Names: immune adjuvant; granulocyte-macrophage colony stimulating factor

SUMMARY:
This research study is evaluating a new type of esophagus cancer vaccine called "Personalized Neoantigen Cancer Vaccine" as a possible treatment for esophagus cancer patients who have completed adjuvant therapy following neoadjuvant therapy and surgical resection. The purpose of the clinical study is evaluating the safety, tolerability and partial efficacy of the personalized neoantigen cancer vaccine in the treatment of resectable esophagus cancer, so as to provide a new personalized therapeutic strategy.

DETAILED DESCRIPTION:
It is known that cancer patients have mutations (changes in genetic material) that are specific to an individual patient and tumor. These mutations can cause the tumor cells to produce proteins that appear very different from the body's own cells. It is possible that these proteins used in a vaccine may induce strong immune responses, which may help the participant's body fight any tumor cells that could cause the cancer to come back in the future. The study will examine the safety of the vaccine when given at several different time points and will examine the participant's blood cells for signs that the vaccine induced an immune response.

ELIGIBILITY:
Inclusion Criteria:

1. Must freely sign informed consent;
2. Aged 18 to 80 years old;
3. Histologically or cytologically confirmed diagnosis of esophagus cancer;
4. ECOG score is 0 or 1;
5. completed Neoadjuvant combined with PD-1 therapy ;Completed surgical resection ;At the same time, standard postoperative treatment was performed 8 ~ 12 weeks of therapy;
6. Must provide all exons of tumor tissue sequencing data, transcriptome sequencing data and the peripheral blood of all exons sequencing data;
7. Completion of imaging records 1 week before personalized immunotherapy, including but not limited to full-body PET-CT and brain MRI,
8. Haematological index： White blood cells ≥ 3500 / MCL; Lymphocytes > 800/ MCL; neutrophils > 1500/ MCL; Platelets > 100000 / MCL; Hemoglobin >10.0g/dL; Total serum bilirubin <1.5× upper limit of normal value (ULN); AST/ALT<2.0 times the upper limit of normal; Serum creatinine <1.5 times the upper limit of normal；
9. Pregnant, lactating women and women of child-bearing age must have a negative pregnancy test within 7 days before entering the group, and short-term have no fertility plan, and are willing to take protective measures (contraception or other birth control methods) before and during the clinical trial;
10. Male patients are willing to take appropriate methods of contraception;
11. Good compliance, able to follow research protocols and follow-up procedures;

Exclusion Criteria:

1. Diagnosed as other malignant tumor;
2. No neoantigen was found in the sequencing data;
3. Patients are unable to tolerate surgery and adjuvant therapy or patients with poor immune system status;
4. There have been bone marrow or stem cell transplants;
5. Received other systemic antitumor agents or systemic glucocorticoids with immunosuppressants;
6. Received other vaccine inoculation 4 weeks before treatment;
7. With HIV, HCV, HBV infection, severe asthma, autoimmune disease,immunodeficiency or treated with immunosuppressive drugs;
8. Uncontrolled complications include, but are not limited to, active infection, symptomatic congestive heart failure, unstable angina pectoris, and arrhythmias;
9. Infected with herpes virus (except those with scabs of more than 4 weeks);
10. Infected with respiratory virus (except those who have recovered for more than 4 weeks);
11. Have severe coronary or cerebrovascular disease, or other conditions considered ineligible by the investigator;
12. Drug abuse. Clinical, psychological or social factor result in affecting informed consent or research implementation;
13. Have a history of drug or vaccine allergies, or people who are allergic to other potential immunotherapies;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
AEs | 1 year
  To evaluate the number of patients with clinical or laboratory adverse events (AEs)
Relapse Free Survival Rate | 1 year
  Proportion of patients who have had surgery for less than 1 year before their first documented relapse

SECONDARY OUTCOMES:
Relapse Free Survival | 3 years
  The time between the patient's completion of surgery and the first recorded relapse
Overall Survival | 3 years
  From the time of the patient's surgery to the time of death
EORTC QLQ-C30 (version 3) | 3 years
  Quality of life questionnaire. All questionnaire responses were transformed linearly to scores from 0 to 100. For functional scores and global QOL, higher scores represent better function and QOL, whereas a higher score for the symptom scales represents more severe symptom.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China